CLINICAL TRIAL: NCT02762825
Title: Novel Cardiac Rehabilitation in Patients Heart Failure and Preserved Ejection Fraction
Acronym: CRpEF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment of eligible patients
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Steven J. Keteyian, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFHS HFpEF HIIT
Record Dates: First submitted 2016-03-22; First posted 2016-05-05 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic

ARMS (2):
- Higher Intensity Interval Training (HIIT) (Experimental)
  Interventions: Behavioral: HIIT
- Moderate Continuous Training (MCT) (Active Comparator)
  Interventions: Behavioral: MCT

INTERVENTIONS:
Behavioral: HIIT — HIIT will consist of 4 min of higher intensity work set at 90% of heart rate reserve, based on peak heart rate from CPX test. Recovery intervals will be 3-4 min in duration and set at 60-70% of heart rate reserve. Resistance training will be performed once per week.
  Arms: Higher Intensity Interval Training (HIIT)
Behavioral: MCT — MCT will consist of aerobic exercise performed 3 times per week for 30 min each session, at an intensity of 60-80% of heart rate reserve, based on peak heart rate from CPX test.
  Arms: Moderate Continuous Training (MCT)

SUMMARY:
Patients with HFpEF suffer from exercise intolerance, increased risk for hospitalization and mortality, and poor QOL. Unlike patients with HFrEF, no drug or device therapies appear to be consistently beneficial in treating these problems. However, increasing evidence suggests that exercise training is effective for both partially reversing exercise intolerance and improving quality of life in these patients. Most such trials to date have been conducted in controlled research setting, versus integrating these patients in to a standard CR program. Also, since functional capacity is related to outcomes in these patients, exercise strategies aimed at further improving fitness are warranted. One such strategy is using higher intensity interval training (HIIT) in the CR setting, a strategy shown to be effective in patients with other types of CVD. This project is designed to test the feasibility of incorporating these patients into the CR setting, and training them using a methodology (i.e., HIIT) already shown to yield (in other patients with CVD) greater gains in fitness when compared to what was achieved using standard MCT alone.

ELIGIBILITY:
Inclusion Criteria:

1. NYHA class II or III symptoms
2. Referred by physician to CR with echocardiographic evidence of HFpEF defined as an ejection fraction ≥ 50 % and moderate to severe (grade II-III) diastolic dysfunction.
3. ≥ 50 years of age
4. Free of orthopedic or other medical problems that would limit participation in CR
5. Peak VO2 on baseline cardiopulmonary exercise test (CPX) < 24 mL/kg/min in men and <21 mL/kg/min in women

Exclusion Criteria:

1. Systolic dysfunction, per ejection fraction < 50%; those with mild (grade I) diastolic dysfunction
2. Initial clinical responses observed during first 3 visits in CR or baseline exercise test that would preclude participation in study over-all (e.g., new onset/troublesome arrhythmia that warrants further investigation) or undergoing HIIT (e.g., claudication, balance issue)
3. Patients with exercise induced angina during CR or CPX testing or ST segment depression representative of myocardial ischemia during CPX testing
4. Pregnant or planning to become pregnant
5. Any patient recently hospitalized for heart failure will have to wait at least 2 weeks before starting CR, or until clinically stable per physician(whichever time period is greater)
6. Atrial fibrillation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen consumption from baseline | Change from baseline at 10-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Keteyian, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States